CLINICAL TRIAL: NCT01084018
Title: Development and Evaluation of a Nursing Virtual Intervention Tailored for Pain After Cardiac Surgery-SOULAGETAVIE
Brief Title: Development and Evaluation of a Nursing Virtual Intervention Tailored for Pain After Cardiac Surgery
Acronym: SOULAGETAVIE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); GRISIIQ (Unknown); FIIC (Unknown); Chaire de recherche sur les nouvelles pratiques de soins infirmiers (Unknown); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: José Côté, CRCHUM
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CE 09.214
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Cardiac Surgery; Pain; Adult; Pain Management
Keywords: acute postoperative pain; nursing intervention
MeSH Terms: conditions — Pain; Agnosia; Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: soulageTAVIE — VITaPaCS consists in a 30 minute-computer-tailored preoperative session, which is animated by a virtual nurse who guides the participant through a learning process about analgesic medication intake, pain communication, and cognitive restructuring. The information and the strategies provided are specifically tailored to the participants' profile, determined by a screening questionnaire, but also by their responses in real-time during the computer session. Two postoperative clinical reinforcements of ten minutes are also provided by the treating nurse based on the flags identified through the preoperative session.

SUMMARY:
The purpose of this project is to develop and evaluate the effects of a computer-tailored intervention targeting pain barriers and catastrophizing in adults having cardiac surgery.

The hypotheses are that in the experimental group, in comparison to the control group, participants will show lower levels of pain, less pain interference in their activities, less attitudinal barriers, and less pain catastrophizing.

A pilot-RCT is privileged to assess the preliminary effects of the intervention on the following outcomes: pain intensity, analgesic consumption, pain interference, barriers and pain catastrophizing.

ELIGIBILITY:
Inclusion Criteria:

* first intention cardiac surgery
* 18 years old or more
* able to fill up questionnaires in french

Exclusion Criteria:

* participation to another psychosocial intervention
* cognitive or psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
pain intensity | 24, 48, 72 hrs, 7 days, 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: José Côté, PhD, Study Director — Centre de Recherche du Centre Hospitalier de l'Université de Montréal; Manon Choinière, PhD, Study Director — Centre de Recherche du Centre Hospitalier de l'Université de Montréal; Géraldine Martorella, PhD (c), Principal Investigator — Université de Montréal
Locations (1):
- Hotel-Dieu (CHUM), Montreal, Quebec, Canada

REFERENCES:
- [Derived] Martorella G, Cote J, Racine M, Choiniere M. Web-based nursing intervention for self-management of pain after cardiac surgery: pilot randomized controlled trial. J Med Internet Res. 2012 Dec 14;14(6):e177. doi: 10.2196/jmir.2070. PMID 23241361